CLINICAL TRIAL: NCT01699568
Title: Stability of Implants With Different Surface Treatment: Randomized Clinical Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Érico Castaldin Fraga Moreira, Master of Science, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: Erico1
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Edentulous Jaws Partially
Keywords: dental implant stability; dental implant surface treatment; resonance frequence analysis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vulcano Actives (Experimental): Implants 4mm x 10mm Vulcano Actives (anodized surface)(AR Torque Vulcano actives), Conexão Sistemas de Prótese, Arujá, Brasil)will be placed on edentulous area in maxilla
  Interventions: Device: RFA
- Porous (Active Comparator): Implants 4mm x 10mm Porous (dual acid-etched surface treatment)(AR Torque Porous, Conexão Sistemas de Prótese, Arujá, Brasil)will be placed on edentulous area in maxilla
  Interventions: Device: RFA

INTERVENTIONS:
Device: RFA — Each week since the surgery the implant stability will be measure with the Osstell mentor to verify the resonance frequence analysis, using the smartpeg number 21
  Other Names: Osstell mentor; resonance frequence analysis

SUMMARY:
Objectives: To compare the stability of implant surface treated by dual acid etching (Porous)and implants with anodized surface (Vulcano) over a period of 16 weeks after installation.

Methods: it will be a clinical study with individuals with missing teeth requiring rehabilitation with dental implants in the maxilla and that fulfill the study inclusion criteria. The research sites will be randomized into two groups: the control group patient's sites receive implant surface treated by dual acid (AR Torque Porous, Connection Implant Systems, Aruja, Brazil) and in the test group implants with anodized surface (AR Torque Vulcano-Actives, Connection Implant Systems, Aruja, Brazil). The evaluation of the stability of the implants will be made over 16 weeks, through resonance frequency analysis with Osstell (Integration Diagnostics AB, Gothenburg, Sweden). Data will be analyzed using descriptive statistics and comparative.

ELIGIBILITY:
Inclusion Criteria:

* patients who have missing teeth in the maxilla,
* over 30 years old and under 60 years old,
* the implant sites with at least 3 months of healing after extraction,
* the implant sites with width and length to installation of an implant of 4 mm x 10 mm.

Exclusion Criteria:

* patients who experience any of the following conditions:
* general contraindications for surgical procedures,
* uncontrolled diabetes,
* severe bruxism or clenching,
* pregnant and lactating women,
* active periodontal disease,
* smoker and user of alcohol or drugs.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Estimated)
Dates: Start 2012-02; Primary Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
implant loss | 4 months
  During the osseointegration, if the implant lose his stability and if it show spin and if the patient have pain, the implant will be removed and the implant will be considered lost

SECONDARY OUTCOMES:
ISQ analysis | 6 months
  Since the implant installation, for the next 8 weeks, and after for the next 4 months, the implant stability will be measure with the Osstell, that will return a number between 0 and 100. This represents the Implant Stability Quotient (ISQ). The difference between the ISQ results will be the secondary outcome measure

CONTACTS AND LOCATIONS:
Overall Officials: Érico Fraga Moreira, Master of Science, Principal Investigator — Student of doctoral program
Locations (1):
- Faculdade de Odontologia da USP, São Paulo, São Paulo, Brazil